CLINICAL TRIAL: NCT03099928
Title: Developing a Positive Psychology Intervention to Improve Health Behaviors in Type 2 Diabetes: Qualitative Research
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director, Massachusetts General Hospital
Other Study IDs: 2014P002578
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualitative Interviews

SUMMARY:
Specific Aim #1 (Qualitative Research): To identify, through qualitative research, deficits in positive affect and associated barriers to completing health behaviors in type 2 DM patients.

Hypothesis: Patients will be able to complete the structured interview, providing information about their own positive emotional states, identifying strategies to enhance positive emotions, linking the presence of positive emotions to better adherence to health-related behaviors, and identifying additional barriers to completing such behaviors.

Specific Aim #2 (Creation of intervention): To use the data gathered from qualitative and quantitative measures to create a positive psychology-based intervention

Hypothesis: Using the information provided in this trial, the investigators will be able to create an intervention, composed of several positive psychology exercises, that is well-matched with a diabetic population and is targeted to the enhancement adherence to health-related behaviors in this population. This intervention will then be ready for next stage testing.

DETAILED DESCRIPTION:
The investigators are proposing to enroll 31 patients with type 2 DM following an outpatient visit to the MGH Diabetes Center or during admission to Ellison 9-11 inpatient units (or sometime in the following 14 days if the participant is not available to complete the interview after consenting for the study).

For these interviews, the investigators will discuss positive emotional states that patients have experienced and talk about ways they might increase these states. The investigators will also touch on health behaviors in which the patient has engaged and whether positive emotions played a role in completing these behaviors. To enhance the accessibility of this project, the investigators chose to allow patients to complete interviews over the phone. Interactions by phone (rather than in-person visits) can allow for patients who are being discharged from the hospital or have no time to complete the interview during a clinic visit.

The investigators will also conduct a follow up phone call 3 months post-hospitalization during which the investigators will collect mood and anxiety data from participants. The purpose of this data will be to better characterize the population, allowing the investigators to better customize the intervention for this population.

There are two study visits (the first of which can be broken into two parts if the participant cannot complete the interview in the hospital after consenting to the study). The first visit will consist of three brief scales of mood and anxiety (Hospital Anxiety and Depression Scale, Positive and Negative Affect Schedule, and Life Orientation Test-Revised) that will take 10 minutes, followed by a 45 minute interview. Participants also will report their race and ethnicity. The second visit will take place 3 months after the initial visit and will be conducted over the phone. This second visit will consist of the same three brief scales of mood and anxiety.

Baseline Data: Baseline information about enrolled subjects will also be obtained from the patients, care providers, the structured assessments of mood and anxiety symptoms as above, and the electronic medical record as required for characterization of our population. This information will include data regarding medical history (history of cardiac illness, diabetes mellitus, hyperlipidemia, and current smoking), current medical variables (admission diagnosis if applicable, HbA1c), medications, length of hospital stay if applicable, and sociodemographic data (age, gender, race/ethnicity, living alone). This information will help the investigators to ensure that the population the investigators recruit is a representative population of patients with type 2 DM.

Qualitative Data: Subjects will undergo an open-ended, one-hour structured interview. The interview will be performed by study staff trained in qualitative research methods by the study PI, Dr. Huffman, using frameworks from Dr. Huffman's prior work. First, subjects will be asked open-ended questions about positive emotional/cognitive experiences. Interviewers will ask about subjects' experience with positive thoughts and feelings recently, and will attempt to elicit both the frequency/intensity of such experiences and the range of such states (e.g., elation vs. optimism). Next, subjects will be asked in an open-ended manner about ideas that they may have to increase the frequency and breadth of their own positive experiences, and then will be asked their opinion about the potential utility of several different existing positive psychology exercises. The interviewers will then inquire about the impact that positive thoughts/feelings may have on our specific diabetes-related health behaviors of interest.

Follow-up 3 Month Phone Call: Three months after discharge from the hospital, a study RA will call subjects to repeat the measures of mood and anxiety completed at baseline (HADS, PANAS, and LOT-R). The investigators will record specific times at enrollment that subjects would prefer to be called (and not to be called) to reduce intrusion on subjects' lives. The investigators will also remind subjects of their upcoming call, in case they need to reschedule. If subjects would rather complete the questions in written form rather than over the phone, the investigators will send them a written packet at the time of each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (21 years and older) admitted to one of the inpatient cardiac units (Ellison 9, 10, or11) at MGH or a current outpatient in the MGH Diabetes Center. Patients must have Type 2 Diabetes (confirmed via medical record and diabetologist/attending physician).
* Suboptimal adherence to health behaviors (diabetic diet, physical activity, medication), as measured by the Medical Outcomes Study Specific Adherence Scale (MOS SAS), as denoted by a score of <15 out of 18.

Exclusion Criteria:

* Cognitive deficits, assessed via a 6-item cognitive screen used to assess appropriate participation of medically-ill patients in research studies.24-26
* Medical conditions precluding interviews, determined in consultation with attending physician or diabetologist.
* Inability to communicate in English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients admitted to three inpatient units or seen at the MGH Diabetes Center.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Qualitative data | Baseline
  Themes related to: Positive psychological states, barriers to health behaviors, relationships between positive states and barriers to health behaviors, and feedback about potential PP exercises

SECONDARY OUTCOMES:
Change in anxiety | Baseline, 3 months
  Measured by the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
Change in depression | Baseline, 3 months
  Measured by the depression subscale of the Hospital Anxiety and Depression Scale (HADS)
Change in positive affective | Baseline, 3 months
  Measured by the Positive and Negative Affect Schedule (PANAS)
Change in optimism | Baseline, 3 months
  Measured by the Life Orientation Test-Revised (LOT-R)

IPD SHARING:
Plan to Share IPD: No